CLINICAL TRIAL: NCT00960089
Title: Evaluation of the Efficacy of Chesson Labs LIQUICURE™ for Treatment of Onychomycosis
Brief Title: Efficacy Study of LIQUICURE™ to Treat Toe Nail Fungus
Acronym: CT001
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chesson Laboratory Associates, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Chesson Labs CT001-01
Record Dates: First submitted 2009-08-14; First posted 2009-08-17 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2016-01

CONDITIONS: Onychomycosis
Keywords: Toenail; Fungus; Onychomycosis; Dermatophyte
MeSH Terms: conditions — Onychomycosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- LIQUICURE (Experimental): Medical Device
  Interventions: Device: LIQUICURE

INTERVENTIONS:
Device: LIQUICURE — Topical treatment, 1 time/day, 5 days/week

SUMMARY:
There is a major clinical need for an inexpensive topically-applied product that can inhibit the growth of the dermatophytes that cause nail fungus. Chesson Labs has developed LIQUICURE with a longer drying/curing time that will allow better nail penetration or adsorption. Though the product may have inherent antimicrobial activity, the product does not contain a drug or antimicrobial agent.

Consistent use of LIQUICURE as described will clear fungal nail infection. Clearing of nail fungal infection is defined by negative dermatophyte culture and visual improvement in nail characteristics within six months, with few, if any product-related adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Nail fungal infection of at least one great toe [per visual assessment, positive KOH preparation, and positive dermatophyte culture]
* Subjects who have target toenail showing 20-65% involvement as judged by the clinical investigator
* 2 mm of clear nail proximally on great toenail / no lunula involvement
* Subject must be physically able to reach toes to clean them and apply product
* Subject is willing to discontinue use of other nail fungus treatment products and nail cosmetic products for duration of this study
* Subject is willing and available to return for study follow up
* Ability of the subject or legal representative to understand and provide signed consent for participating in the study
* Negative urine pregnancy test for women of child bearing age
* Females must be post menopausal or must agree to use approved contraceptives (actions, devices or medications to prevent or reduce the likelihood of pregnancy) throughout the study (Note: abstinence is NOT an accepted form of contraception)

Exclusion Criteria:

* Known hypersensitivity or allergy to the product materials
* Negative KOH preparation or dermatophyte culture
* Thickness of nail greater than 3 mm
* Enrollment in another investigational drug or product protocol that would interfere with this study
* Continuation or use of other topical or pharmaceutical treatments for the condition; a wash-out period of at least four weeks after discontinuation of a topical product or 180 days after discontinuation of an oral product for treatment of nail fungus is required
* Chronic disease, including: diabetes, psoriasis, immune deficiency, severe foot injury, chronic vascular disease or any other condition that would decrease circulation to the extremities at the discretion of the investigator Pregnant or nursing females
* Investigators, Chesson personnel, or Chesson Scientific Advisory Board members or their immediate family

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2008-07; Primary Completion 2010-04 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Freedom from major product-related adverse events for the duration of the feasibility phase. | Six months
Clearance of fungal nail infection defined by negative culture and improvement in visual nail characteristics | Six months

SECONDARY OUTCOMES:
Time to clearance of infection | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Beth Goldstein, MD, Principal Investigator — Central Dermatology
Locations (4):
- United States (4):
  - Triangle Medical Research Associates, Cary, North Carolina
  - Central Dermatology Center, Chapel Hill, North Carolina
  - Wake Research Associates, Raleigh, North Carolina
  - Crescent Medical Research, Salisbury, North Carolina